CLINICAL TRIAL: NCT05498051
Title: A Pilot Study to Assess the Safety and Feasibility of Fluorescent Sentinel Lymph Node Identification in Colon Carcinoma Using Submucosal Bevacizumab-800CW.
Brief Title: Fluorescent Sentinel Lymph Node Identification in Colon Carcinoma Using Submucosal Bevacizumab-800CW.
Acronym: IBIZA-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meander Medical Center (Other)
Responsible Party: Principal Investigator, Esther Consten, prof. dr., Meander Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21.116; 2021-006700-32 (EudraCT Number)
Record Dates: First submitted 2022-07-20; First posted 2022-08-11 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Colonic Neoplasms; Sentinel Lymph Node; Fluorescence; Colorectal Neoplasms
Keywords: Sentinel lymph node; Colon cancer; Fluorescence; bevacizumab-800CW; bevacizumab-IRdye
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single-centre, open-label, non-randomized cohort safety and feasibility study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sentinel lymph node detection after submucosal bevacizumab-800CW injection (Experimental): Therefore this prospective study aims to assess the safety and feasibility of lymph node identification using bevacizumab-800CW in patients with cT1-3N0-2 tumours, using peritumoral submucosal injections.
  Interventions: Procedure: Sentinel lymph node identification

INTERVENTIONS:
Procedure: Sentinel lymph node identification — Therefore this prospective study aims to assess the safety and feasibility of lymph node identification using bevacizumab-800CW in patients with cT1-3N0-2 tumours, using peritumoral submucosal injections.
  Other Names: SLN

SUMMARY:
This prospective study aims to assess the safety and feasibility of lymph node identification using bevacizumab-800CW in patients with cT1-3N0-2 tumours, using peritumoral submucosal injections

DETAILED DESCRIPTION:
The current gold standard for the treatment of colon carcinoma consists of the surgical en-bloc resection of the colonic segment including the adjacent mesocolon containing the draining lymph nodes. Analysis of these lymph nodes is important, since lymph node status is one of the most important prognostic factors determining the use of adjuvant chemotherapy. Although patients with tumour stage I and II do not have lymph node metastases, 15-20% develop recurrent disease. Several studies suggest that ultrastaging techniques such as immunohistochemistry (IHC) or reverse transcriptase polymerase chain reaction (RT-PCR) using multilevel slicing results in upstaging of 14-18% of patients, due to newly found (micro)metastasis. Furthermore, several studies indicate that these micrometastases are correlated with a significantly poorer prognosis, subsequently suggesting that this subgroup of patients might benefit of adjuvant chemotherapy. Therefore, the most recent Dutch guidelines advice the use of adjuvant chemotherapy in this "upstaged" group, although evidence is still lacking.

However, ultrastaging techniques are labour-intensive and costly, and therefore not suitable for analyses of all lymph nodes that have been collected during segmental colectomy. Sentinel lymph node (SLN) identification in colon carcinoma has been proposed to overcome this problem by identifying the first order draining lymph node(s) of the tumour, which have the highest chance of containing metastatic tumour cells. Several studies aimed at SLN identification in colon carcinoma have been published, however, early studies using radio-guided or blue-dye guided SLN identification, showed relatively high rates of false negatives with consequent low sensitivity rates. Since mesocolon is rather fatty tissue, visualization of conventional dyes is difficult. Indocyanine green (ICG), which can be visualized using near infrared (NIR), has been put forward since it is known to penetrate relatively deep into living tissue.

Nevertheless, results of SLN identification using ICG remain unsatisfying with high false-negative rates and low sensitivity. Most likely this is due to the fact that these studies also included large cT3-cT4 tumours and patients with massive lymph node involvement. Which are factors known to interfere with lymph drainage patterns. Furthermore, subserosal injections were frequently used, while it is suggested that submucosal injections might result in better sensitivity of the procedure. In the FLUOR-SLN-ICG pilot study, we successfully conducted SLN identification in patients with ICG.

Recently, more research is conducted in tumour-targeted tracers as they have many advantages compared to ICG. For example, tumour-targeted tracers can be preoperatively administered which aid logistics, binds to tumour and metastases, thus allowing more time for uptake in patients with larger tumours and lymph node metastases. These properties may result in increased accuracy and would be more broadly applicable compared to ICG. Furthermore, tumour-targeted tracers can also be administrated intravenously and potentially identify lymph node metastases without having to perform a colonoscopy. However, administration via colonoscopy of tumour-targeted tracers for the detection of lymph node metastases in colon carcinoma has not been performed yet, and intravenous administration would be a step after administration via colonoscopy.

Therefore this prospective study aims to assess the safety and feasibility of lymph node identification using bevacizumab-800CW in patients with cT1-3N0-2 tumours, using peritumoral submucosal injections.

ELIGIBILITY:
Inclusion Criteria:

* Oral and written informed consent (IC)
* Aged 18 years and older
* Patients with pathologically confirmed and/or suspected cT1-3N0-2M0 colon carcinoma.

Exclusion Criteria:

* Distant metastasis
* Suspicion of cT4 disease based on pre-operative assessment
* Metastatic or T4 disease discovered during intraoperative staging
* Pregnancy, lactation or a planned pregnancy during the course of the study
* Previous colon surgery, excluding appendectomy.
* Contra-indication for laparoscopic/robotic surgery
* Inadequately controlled hypertension with or without current antihypertensive medication.
* Within 6 months prior to inclusion: myocardial infarction, TIA, CVA, pulmonary embolism, unstable angina pectoris, or uncontrolled chronic hepatic failure.
* Regarding Bevacizumab: Hypersensitivity to Chinese Hamster Ovary (CHO) cell products or other recombinant human or humanised antibodies. Or an allergy for it's components (Trehalose dehydrate, sodium phosphate, polysorbate 20, water for injections)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Identification rate of SLN(s) or lymph node metastases | During surgery
  Defined as the number of patients in which a SLN or lymph node metastases were detected due to fluorescence during surgery and/or pathology assessment divided by the total number of procedures.
  We conclude that the study is a feasible if:
  * We are to detect fluorescence in lymph nodes in 3 out of 5 patients (regardless of the presence of metastases)
  * And/or we are able to detect lymph node metastases with fluorescence, or if fluorescence is higher in lymph node metastases compared to tumour-negative lymph nodes.
Safety of SLN identification | Measured till 90 days after surgery
  The rate of adverse events related to bevacizumab-800CW (injection) will be measured. This is defined as the number of adverse events related towards bevacizumab-800CW/total number of procedures.

SECONDARY OUTCOMES:
Amount of fluorescence in lymph node metastases compared to lymph node without metastases | 3 months (after fluorescence measurement)
  Fluorescence measured in the Oddysey flatbed scanner
false-negative SLNs | 3 months (after pathological examination)
  The SLNs are negative whereas the non-sentinel nodes (NSNs) were positive (number).
true-negative SLNs | 3 months (after pathological examination)
  Both the SLNs and NSNs are negative (number).
sensitivity | 3 months (after pathological examination)
  The number of patients with a positive SLN / the total number of node positive patients (n, %).
upstaged patients | 3 months (after pathological examination)
  The number of patients with SLNs positive for micro- or macrometastases by serial slicing and IHC / the number of patients who were node negative by H&E examination (n, %).
aberrant lymph node status | 3 months (after pathological examination)
  The number of patients with aberrant lymph nodes, and the status of these lymph nodes considering micro- or macrometastases.
accuracy | 3 months (after pathological examination)
  (The total number of patients with a positive SLN + the number of patients with a true-negative SLN) / number of patients with an identified SLN (n, %).
negative predictive value | 3 months (after pathological examination)
  The number of true negative SLNs / (true negative + false negative SLNs).
number of SLNs identified | 3 months (after pathological examination)
  Number of SLN identified (number).

CONTACTS AND LOCATIONS:
Overall Officials: Esther Consten, prof. dr., Principal Investigator — Meander Medisch Centrum
Locations (1):
- Meander Medisch Centrum, Amersfoort, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided